CLINICAL TRIAL: NCT05344027
Title: The Impact of Mitotane Therapy on Serum Free Proteins in Patients With Adrenocortical Carcinoma
Acronym: MitoS-FP
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GafREC-Endo202
Record Dates: First submitted 2022-04-11; First posted 2022-04-25 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Adrenocortical Carcinoma
Keywords: mitotane; adrenocortical carcinoma; ACC; serum free proteins; cortisol binding globulin; thyroid binding globulin
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Mitotane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ACC on mitotane: Individuals in this group were under care by the Endocrinology Team with a diagnosis of an ACC and on mitotane. These individuals were further divided into 3 groups, depending on whether they had a mitotane plasma concentration, within (14-20mg/L), above or below the therapeutic concentration range.
  Interventions: Drug: Mitotane
- Adrenal neoplasm without mitotane: Individuals within this category had an adrenal neoplasm and were not being treated with mitotane therapy.
- Pregnant group: Individuals did not have an adrenal neoplasm during this period, nor were they being treated with mitotane. These were healthy pregnant females, who were under the care at KCL during their pregnancy.

INTERVENTIONS:
Drug: Mitotane — Individuals within the intervention group were on mitotane therapy as part of their ACC treatment.
  Groups: ACC on mitotane

SUMMARY:
This work will evaluate the effects of mitotane treatment on serum protein concentrations in patients treated for ACC with mitotane therapy and compare them to patients with an adrenal neoplasm and pregnant cohort. All of the individuals were treated at King's Hospital between April 2019 and June 2020. Proteins which will be evaluated during this study, include CBG and TBG.

DETAILED DESCRIPTION:
Background: Adrenocortical Carcinoma (ACC) is a rare malignancy of the adrenal cortex. The annual incidence of ACC is thought to be between 0.5-2.0 cases per million. Adjunctive therapy with mitotane may be offered post- surgically to minimise risk of recurrence.

Aims: Evaluate the effects of mitotane treatment on serum protein concentrations in patients treated for ACC with mitotane therapy and compare to patients with an adrenal neoplasm and a pregnant cohort. Patients were treated at King's Hospital between April 2019 and June 2020.

Methods: Cortisol, TFT's ACTH, CBG, TBG and gonadotrophins will be measured during the same venepuncture using serum samples. SPSS v27 and GraphPad Prism v9.3.1 will be used for analysis and illustrations. Thirty-five patients will be included, within ACC with mitotane, adrenal neoplasm or pregnant groups. Data will be tested for normality, described as Mean± SD, compared using paired sample t-test with 5% p-value for significance and 95% confidence interval (CI).

ELIGIBILITY:
Inclusion Criteria: An individual being investigated for a malignant neoplasm treated with mitotane or matched number of patients with adrenal neoplasm not treated with mitotane under the Endocrinology team or a matched cohort of pregnant women.

Patients included in the analysis were seen in the period between April of 2019 and June 2020 at King's College Hospital NHS Foundation Trust.

-

Exclusion Criteria:

* Patients not investigated for a malignant neoplasm/ adrenal neoplasm under the Endocrinology team or were a matched cohort of pregnant women at King's College Hospital NHS Foundation Trust during the period Someone under the age of 18

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 13 patients with an ACC on mitotane therapy will be investigated. Median age of the ACC and mitotane group: 63.0 (IQR: 46, 72.5) 22% of the studied population were Caucasian white, 14.3% Southeast Asian, 11.4% Black Afro-Caribbean, 2.9% other and 2.9% missing. 6 (46.2%) of the patients with an ACC and on mitotane were male, and 7 (53.8%) were female. 6 (46.2%) individuals with an ACC and on mitotane had a stage of III and 7 (53.8%) had stage IV (according to the AJCC and ENSAT staging system).
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Examine the effect of mitotane therapy on serum thyroid and cortisol binding proteins in patients with ACC | April 2019-June 2020
  The primary objective of this project is to determine the effects of mitotane therapy on serum thyroid binding and cortisol binding protein concentrations in patients with adrenocortical carcinoma and compare concentrations of the same binding proteins in patients with adrenal neoplasms not on treatment with mitotane and to a cohort of pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kerkhofs TM, Verhoeven RH, Van der Zwan JM, Dieleman J, Kerstens MN, Links TP, Van de Poll-Franse LV, Haak HR. Adrenocortical carcinoma: a population-based study on incidence and survival in the Netherlands since 1993. Eur J Cancer. 2013 Jul;49(11):2579-86. doi: 10.1016/j.ejca.2013.02.034. Epub 2013 Apr 3. PMID 23561851
- [Background] Scollo C, Russo M, Trovato MA, Sambataro D, Giuffrida D, Manusia M, Sapuppo G, Malandrino P, Vigneri R, Pellegriti G. Prognostic Factors for Adrenocortical Carcinoma Outcomes. Front Endocrinol (Lausanne). 2016 Jul 25;7:99. doi: 10.3389/fendo.2016.00099. eCollection 2016. PMID 27504106
- [Background] Alexandraki KI, Kaltsas GA, le Roux CW, Fassnacht M, Ajodha S, Christ-Crain M, Akker SA, Drake WM, Edwards R, Allolio B, Grossman AB. Assessment of serum-free cortisol levels in patients with adrenocortical carcinoma treated with mitotane: a pilot study. Clin Endocrinol (Oxf). 2010 Mar;72(3):305-11. doi: 10.1111/j.1365-2265.2009.03631.x. Epub 2009 May 16. PMID 19473175
- [Background] Russo M, Scollo C, Pellegriti G, Cotta OR, Squatrito S, Frasca F, Cannavo S, Gullo D. Mitotane treatment in patients with adrenocortical cancer causes central hypothyroidism. Clin Endocrinol (Oxf). 2016 Apr;84(4):614-9. doi: 10.1111/cen.12868. Epub 2015 Aug 18. PMID 26221968
- [Background] Fassnacht M, Allolio B. Clinical management of adrenocortical carcinoma. Best Pract Res Clin Endocrinol Metab. 2009 Apr;23(2):273-89. doi: 10.1016/j.beem.2008.10.008. PMID 19500769
- [Background] Allolio B, Fassnacht M. Clinical review: Adrenocortical carcinoma: clinical update. J Clin Endocrinol Metab. 2006 Jun;91(6):2027-37. doi: 10.1210/jc.2005-2639. Epub 2006 Mar 21. PMID 16551738
- [Background] van Erp NP, Guchelaar HJ, Ploeger BA, Romijn JA, Hartigh Jd, Gelderblom H. Mitotane has a strong and a durable inducing effect on CYP3A4 activity. Eur J Endocrinol. 2011 Apr;164(4):621-6. doi: 10.1530/EJE-10-0956. Epub 2011 Jan 10. PMID 21220434
- [Background] Fassnacht M, Assie G, Baudin E, Eisenhofer G, de la Fouchardiere C, Haak HR, de Krijger R, Porpiglia F, Terzolo M, Berruti A; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Adrenocortical carcinomas and malignant phaeochromocytomas: ESMO-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Nov;31(11):1476-1490. doi: 10.1016/j.annonc.2020.08.2099. Epub 2020 Aug 27. No abstract available. PMID 32861807
- [Background] Sada A, Glasgow AE, Lyden ML, Dy BM, Foster TR, Habermann EB, Bancos I, McKenzie TJ. Informing therapeutic lymphadenectomy: Location of regional metastatic lymph nodes in adrenocortical carcinoma. Am J Surg. 2022 Jun;223(6):1042-1045. doi: 10.1016/j.amjsurg.2021.10.014. Epub 2021 Oct 19. PMID 34696848
- [Background] Lehmann TP, Wrzesinski T, Jagodzinski PP. The effect of mitotane on viability, steroidogenesis and gene expression in NCI-H295R adrenocortical cells. Mol Med Rep. 2013 Mar;7(3):893-900. doi: 10.3892/mmr.2012.1244. Epub 2012 Dec 18. PMID 23254310
- [Background] Tran TB, Liou D, Menon VG, Nissen NN. Surgical management of advanced adrenocortical carcinoma: a 21-year population-based analysis. Am Surg. 2013 Oct;79(10):1115-8. PMID 24160811
- [Background] van Seters AP, Moolenaar AJ. Mitotane increases the blood levels of hormone-binding proteins. Acta Endocrinol (Copenh). 1991 May;124(5):526-33. doi: 10.1530/acta.0.1240526. PMID 1903011
- [Result] Daffara F, De Francia S, Reimondo G, Zaggia B, Aroasio E, Porpiglia F, Volante M, Termine A, Di Carlo F, Dogliotti L, Angeli A, Berruti A, Terzolo M. Prospective evaluation of mitotane toxicity in adrenocortical cancer patients treated adjuvantly. Endocr Relat Cancer. 2008 Dec;15(4):1043-53. doi: 10.1677/ERC-08-0103. Epub 2008 Sep 29. PMID 18824557
- [Result] Fassnacht M, Dekkers OM, Else T, Baudin E, Berruti A, de Krijger R, Haak HR, Mihai R, Assie G, Terzolo M. European Society of Endocrinology Clinical Practice Guidelines on the management of adrenocortical carcinoma in adults, in collaboration with the European Network for the Study of Adrenal Tumors. Eur J Endocrinol. 2018 Oct 1;179(4):G1-G46. doi: 10.1530/EJE-18-0608. PMID 30299884
- [Result] Fassnacht M, Terzolo M, Allolio B, Baudin E, Haak H, Berruti A, Welin S, Schade-Brittinger C, Lacroix A, Jarzab B, Sorbye H, Torpy DJ, Stepan V, Schteingart DE, Arlt W, Kroiss M, Leboulleux S, Sperone P, Sundin A, Hermsen I, Hahner S, Willenberg HS, Tabarin A, Quinkler M, de la Fouchardiere C, Schlumberger M, Mantero F, Weismann D, Beuschlein F, Gelderblom H, Wilmink H, Sender M, Edgerly M, Kenn W, Fojo T, Muller HH, Skogseid B; FIRM-ACT Study Group. Combination chemotherapy in advanced adrenocortical carcinoma. N Engl J Med. 2012 Jun 7;366(23):2189-97. doi: 10.1056/NEJMoa1200966. Epub 2012 May 2. PMID 22551107
- See also: Adrenal Carcinoma Risk Factors — https://moffitt.org/cancers/adrenal-cancer/diagnosis/risk-factors/
- See also: Lysodren (mitotane) dosing, indications, interactions, adverse effects, and more. — https://reference.medscape.com/drug/lysodren-mitotane-342258#10
- See also: Drug Metabolism — https://www.medsafe.govt.nz/profs/puarticles/march2014drugmetabolismcytochromep4503a4.htm
- See also: Dehydroepiandrosterone and Dehydroepiandrosterone Sulfate - Health Encyclopedia — http://www.urmc.rochester.edu/encyclopedia/content.aspx?contenttypeid=167&contentid=dhea
- See also: Cortisol | South Tees Hospitals NHS Foundation Trust — http://www.southtees.nhs.uk/services/pathology/tests/cortisol/
- See also: Adrenal Cancer Stages — http://www.cancer.org/cancer/adrenal-cancer/detection-diagnosis-staging/staging.html